CLINICAL TRIAL: NCT02803645
Title: Clinical Significance of Antiphospholipid Antibodies in Healthy Subjects: Study of Their Association With Cardiovascular Risk Factors, Markers of Arterial Inflammation and Markers of Oxidative Stress
Brief Title: Clinical Significance of Antiphospholipid Antibodies in Healthy Subjects
Acronym: SAPL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PHRCIR05-DR-SALLE
Record Dates: First submitted 2016-06-09; First posted 2016-06-17 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Antiphospholipid Antibodies
Keywords: healthy subjects; cardiovascular risk factors; markers of arterial inflammation; markers of oxidative stress
MeSH Terms: interventions — Blood Specimen Collection

ARMS (1):
- healthy (Experimental): blood sample
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample

SUMMARY:
Antiphospholipid (APL) antibodies are a heterogeneous family of auto-antibodies, predominantly represented by anticardiolipin (ACL) antibodies and lupus anticoagulant (LA). Antiphospholipid syndrome (APS) is defined as the presence of APL associated with venous and/or arterial thrombosis or repeated foetal loss. APS may be either primary or secondary to an autoimmune disease, mainly systemic lupus erythematosus (SLE). However, other than in the context of APS, APL can also be observed in various clinical situations and in healthy subjects. Published studies have reported a variable prevalence of APL in healthy subjects, essentially ACL and/or LA, and their clinical significance currently remains unclear.

Several studies have highlighted the link between APL and atherosclerosis. It therefore appears interesting to more specifically study the association between the presence of APL and the presence of cardiovascular risk factors in a population of healthy subjects. Atherosclerosis is currently considered to be a chronic inflammatory disease arising from a complex interaction between atherogenic plasma factors and cells of the arterial wall. Several inflammatory markers are now known to be associated with cardiovascular risk. Lipid peroxidation also plays a major role during the atherogenesis process. It will therefore also be important to correlate APL with markers of vascular inflammation and markers of oxidative stress.

A prospective case-control study will therefore be conducted on 1,500 healthy blood donors. Subjects screened APL-positive will be compared to APL-negative subjects in terms of cardiovascular risk factors (cardiovascular risk per se, the presence of cardiovascular disease will not be studied). In the context of a blood donation, all subjects wishing to participate in this study will attend a medical interview and a clinical examination during which various data will be collected, mainly the presence of cardiovascular risk factors. A blood sample will also be taken to assay the various laboratory markers studied.

This study should provide a better understanding of the role of APL in healthy subjects and more clearly specify their possible link with atherosclerosis in this population.

ELIGIBILITY:
Inclusion Criteria:

* healthy blood donors

Exclusion Criteria:

* contraindication to blood donation

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1282 (Actual)
Dates: Start 2007-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
antiphospholipid (APL) antibodies | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Valéry SALLE, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France